CLINICAL TRIAL: NCT06551116
Title: QuantifyHER: Quantitative Immunofluorescence and/or RT-qPCR for Measuring HER2 in HER2-low Metastatic Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); Danaher Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: UPCC 09124; 855924 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2024-07-29; First posted 2024-08-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-05

CONDITIONS: HER2-positive Metastatic Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients can consent to having the study team retain and utilize biospecimens for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HER2 Assay: Analysis of HER2 expression via QIF and mRNA assays
  Interventions: Diagnostic Test: CE-10-IVD

INTERVENTIONS:
Diagnostic Test: CE-10-IVD — Leftover tumor tissue from a routine biopsy will be sent for analysis.

SUMMARY:
This study will assess whether a quantitative, HER2 assay can accurately and reliably discriminate between responders and non-responders among patients with HER2 IHCI+ metastatic breast cancer who are receiving T-Dxd.

ELIGIBILITY:
Inclusion Criteria:

* Women and men age > 18 years
* Metastatic breast cancer, histologically- confirmed. Any estrogen receptor (ER) status is allowed. ER status will be determined by local laboratory assessment utilizing ASCO/CAP guidelines.
* Primary and/or metastatic tumor with 1+ level of expression of HER2 by immunohistochemistry as determined by local laboratory assessment utilizing ASCO/CAP guidelines.
* Measurable disease by cross-sectional imaging at the start of treatment. Patients with measurable bone-only disease or active brain metastases are eligible.
* Archival tissue available for biomarker assessment. One specimen should be the most recent metastatic biopsy. If HER2 1+ status was determined on a different specimen (either primary or metastatic tissue), that specimen is also required. Samples obtained from bone metastases that were processed via decalcification methods are not eligible.
* Intention to initiate therapy with T-DXd (Enhertu) at FDA-approved dose and schedule as next line of therapy. If T-DXd was already initiated, patients must be registered within 30 days of initiation.
* Ability to provide informed consent

Exclusion Criteria:

* Concurrent Her2-overexpressing metastatic breast cancer (as confirmed by a metastatic biopsy with IHC 3+ or IHC 2+ with FISH amplified as per standard ASCO/CAP guidelines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2 IHC1+ metastatic breast cancer, histologically confirmed
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Real-World Objective Response Rate | from date of first dose of T-DXd to date of last dose of T-DXd for each. Up to 100 months
  Association between quantitative HER2 expression (as a continuous variable) and real-world objective response rate

SECONDARY OUTCOMES:
Real-World Progression Free Survival | from date of first dose of T-DXd to date of last dose of T-DXd for each.Up to 100 months
  Association between quantitative HER2 expression (as a continuous variable) and real world Progression Free Survival
Real-World Progression Free Survival and Objective Response Rate by estrogen receptor expression | from date of first dose of T-DXd to date of last dose of T-DXd for each. Up to 100 months
  Association between HER2 expression by quantitative immunofluorescence and mRNA in HER2 IHC 1+ tumors and both rwORR and rwPFS, stratified by mRNA ER expression
Threshold for HER2 QIF and/or mRNA levels | from date of first dose of T-DXd to date of last dose of T-DXd for each. Up to 100 months
  cut-off value for HER2 QIF, mRNA and the combination below which patients will not respond to T-DXd."
Association between combined mRNA + QIF and real-world Objective Response Rate | from date of first dose of T-DXd to date of last dose of T-DXd for each. Up to 100 months
  Comparison, based on rwORR, of a linear combination of HER2 QIF and mRNA, versus either alone in ability to discriminate T-DXd responders from non- responders

CONTACTS AND LOCATIONS:
Overall Officials: Angela DeMichele, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (36):
- United States (36):
  - University of California San Francisco Medical Center, San Francisco, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center, Fairfield, Connecticut
  - Smilow Cancer Hospital at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center, Guilford, Connecticut
  - Smilow Cancer Hospital at Saint Francis, Hartford, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, New Haven, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Georgetown University - Lombardi CCC, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - University of Chicago Medicine Northwest Indiana, Crown Point, Indiana
  - John's Hopkins Hospital, Baltimore, Maryland
  - Montefiore Einstein Medical Center, The Bronx, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UPMC Hillman CC, Pittsburgh, Pennsylvania
  - Smilow Cancer Hospital Care Center, Westerly, Rhode Island
  - Ben Taub General Hospital, Houston, Texas
  - MD Anderson Cancer center, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - MD Anderson Cancer center, League City, Texas
  - MD Anderson Cancer Center, Sugar Land, Texas
  - MD Anderson Cancer center, Woodland, Texas
  - University of Washington - Fred Hutchinson Cancer Center, Seattle, Washington

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT06551116/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT06551116/ICF_001.pdf